CLINICAL TRIAL: NCT00651859
Title: Safety and Efficacy Study of Bimatoprost in Ethnically Japanese Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-024
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): Bimatoprost 0.01% Ophthalmic Solution
  Interventions: Drug: Bimatoprost 0.01% Ophthalmic Solution
- 2 (Experimental): Bimatoprost 0.03% Ophthalmic Solution
  Interventions: Drug: Bimatoprost 0.03% Ophthalmic Solution
- 3 (Placebo Comparator): Bimatoprost Vehicle Ophthalmic Solution
  Interventions: Drug: Bimatoprost Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Bimatoprost 0.01% Ophthalmic Solution — Bimatoprost 0.01% ophthalmic solution 1 drop instilled in each eye once daily in the evening between 19:00 and 21:00
  Arms: 1
Drug: Bimatoprost 0.03% Ophthalmic Solution — Bimatoprost 0.03% ophthalmic solution 1 drop instilled in each eye once daily in the evening between 19:00 and 21:00
  Other Names: LUMIGAN®
  Arms: 2
Drug: Bimatoprost Vehicle Ophthalmic Solution — Bimatoprost vehicle ophthalmic solution 1 drop instilled in each eye once daily in the evening between 19:00 and 21:00
  Arms: 3

SUMMARY:
This study evaluates the safety and efficacy of once-daily bimatoprost 0.03% and 0.01% ophthalmic solutions compared with once-daily administered bimatoprost vehicle ophthalmic solution for 2 weeks in ethnically Japanese patients with open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Ethnically Japanese patients with glaucoma or ocular hypertension in each eye who require IOP-lowering therapy in both eyes

Exclusion Criteria:

* Uncontrolled systemic disease
* Use of bimatoprost or an ocular prostaglandin (eg, latanoprost, travoprost) within 6 weeks prior to baseline (Day 0)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2002-11; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | Day 14

SECONDARY OUTCOMES:
IOP | Days 2 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Francisco, California, United States

REFERENCES:
- See also: Link to Clinical Trial Results — http://www.allerganclinicaltrials.com